CLINICAL TRIAL: NCT04868032
Title: Gaining Optimism After Weight Loss Surgery (GOALS) II: Randomized Controlled Trial of a Positive Psychology-based Intervention to Increase Physical Activity After Bariatric Surgery
Brief Title: Gaining Optimism After Weight Loss Surgery (GOALS) II
Acronym: GOALS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Emily Feig, Ph.D., Instructor in Psychology, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021P001006b; 5K23HL148017 (NIH)
Record Dates: First submitted 2021-04-28; First posted 2021-04-30 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Bariatric Surgery
Keywords: Positive Psychology; Motivational Interviewing; Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: A research assistant blinded to study condition will conduct follow-up assessment visits.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Positive Psychology-Motivational Interviewing Intervention (Experimental): Participants will receive a written treatment manual with detailed information about each topic. The intervention consists of 10 weekly phone sessions (30 minutes each). Each session includes a new psychological skill designed to increase positive emotions experienced during physical activity, a motivational skill designed to boost physical activity, and setting a physical activity goal for the next week using information from the Fitbit. A motivational interviewing approach will be used for all topics.
  Interventions: Behavioral: Positive Psychology-Motivational Interviewing
- Physical Activity Education Control (Active Comparator): Participants randomized to this condition will be provided with a Fitbit, and will be mailed educational materials about physical activity at 4 time points throughout the intervention period. They will not receive a manual or phone calls with an interventionist.
  Interventions: Behavioral: Physical Activity Education Control

INTERVENTIONS:
Behavioral: Positive Psychology-Motivational Interviewing — Participants will receive a written treatment manual with detailed information about each topic. The intervention consists of 10 weekly phone sessions (30 minutes each). Each session includes a new psychological skill designed to increase positive emotions experienced during physical activity, a motivational skill designed to boost physical activity, and setting a physical activity goal for the next week using information from the Fitbit. A motivational interviewing approach will be used for all topics.
  Arms: Positive Psychology-Motivational Interviewing Intervention
Behavioral: Physical Activity Education Control — Participants randomized to this condition will be provided with a Fitbit, and will be mailed educational materials about physical activity at 4 time points throughout the intervention period. They will not receive a manual or phone calls with an interventionist.
  Arms: Physical Activity Education Control

SUMMARY:
This randomized controlled trial examines the feasibility, acceptability, and preliminary impact of an adapted positive psychology-motivational interviewing (PP-MI) intervention for physical activity among patients who have recently undergone bariatric surgery compared to an enhanced usual care control.

DETAILED DESCRIPTION:
This study will test a positive psychology-motivational interviewing (PP-MI) intervention for physical activity promotion in patients who have had bariatric surgery within the past 6-12 months compared to an enhanced usual care control. The investigators will enroll and randomize 58 participants. Study participation includes attending four study visits (two at baseline, one at 10 weeks, and one at 24 weeks). Participants will be randomized either to a 10-week physical activity intervention that includes once-weekly phone calls, a written manual, and a Fitbit activity tracker, or provision of the Fitbit alone. Primary outcomes include the feasibility and acceptability of the intervention. Secondary outcomes include changes in physical activity and other psychological, behavioral, and physiological outcomes at 10 and 24 weeks compared to the control.

ELIGIBILITY:
Inclusion Criteria:

* Adult (age 18+)
* History of bariatric surgery (gastric bypass or sleeve gastrectomy) at one of two academic medical centers within the past 6-12 months
* Interest in increasing physical activity
* Low physical activity, defined as <200 minutes/week self-reported moderate- to-vigorous physical activity
* Access to telephone for study sessions
* Able to read and speak English

Exclusion Criteria:

* Cognitive deficits precluding participation or informed consent
* Illness likely to lead to death in the next 6 months
* Inability to be physically active (e.g., severe arthritis)
* Participation in another program targeting physical activity besides their standard offerings at the surgery center.
* Severe psychiatric condition limiting ability to participate (e.g., psychosis, active substance use disorder)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2025-02-03 (Actual); Study Completion 2025-06-03 (Actual)

PRIMARY OUTCOMES:
Number of intervention sessions completed | 10 weeks
  Feasibility will be measured by examining the number of completed intervention sessions for individuals randomized to the PP-MI intervention. The intervention will be considered feasible if at least 7/10 sessions are completed, on average.
Ease and utility of intervention sessions | 10 weeks
  Acceptability will be measured with ratings of ease and utility after each exercise, measured on a 10-point Likert scale (1=very difficult/not at all helpful, 10=very easy/very helpful). The intervention will be considered acceptable if average ease and utility ratings are at least 7/10.

SECONDARY OUTCOMES:
Change in Moderate to Vigorous Physical Activity (MVPA) | Baseline, 10-Week Follow-Up, 24-Week Follow-Up
  We will use ActiGraph GT3X-BT accelerometers to objectively measure physical activity for 1 week at each assessment. MVPA will be measured in minutes/day.
Change in Steps | Baseline, 10-Week Follow-Up, 24-Week Follow-Up
  Measured by Actigraph accelerometer, in number of steps per day.
Change in Light Physical Activity | Baseline, 10-Week Follow-Up, 24-Week Follow-Up
  Measured by Actigraph accelerometer, in minutes per day.
Change in Sedentary Time | Baseline, 10-Week Follow-Up, 24-Week Follow-Up
  Measured by Actigraph accelerometer, in minutes per day.
Change in Positive Affect | Baseline, 10-Week Follow-Up, 24-Week Follow-Up
  The positive affect items on the Positive and Negative Affect Schedule (PANAS), a well-validated scale used in other intervention trials and in patients with medical illnesses, will be used to measure positive affect (Range: 10-50). Higher scores indicate higher levels of positive affect.
Change in Negative Affect | Baseline, 10-Week Follow-Up, 24-Week Follow-Up
  The negative affect items on the Positive and Negative Affect Schedule (PANAS), a well-validated scale used in other intervention trials and in patients with medical illnesses, will be used to measure negative affect (Range: 10-50). Higher scores indicate higher levels of negative affect.
Change in Optimism | Baseline, 10-Week Follow-Up, 24-Week Follow-Up
  The Life Orientation Test-Revised (LOT-R) is a well-validated 6-item instrument used to measure dispositional optimism (Range: 0-24). Higher scores indicate higher levels of optimism.
Change in Depressive symptoms | Baseline, 10-Week Follow-Up, 24-Week Follow-Up
  The Hospital Anxiety and Depression Scale (HADS)-depression subscale will be used to measure depression. This is a well-validated scale with few somatic symptom items that can confound mood/anxiety assessment in medically-ill patients (Range: 0-21). Higher scores indicate higher levels of depression.
Change in Anxiety | Baseline, 10-Week Follow-Up, 24-Week Follow-Up
  The Hospital Anxiety and Depression Scale (HADS)-anxiety subscale will be used to measure anxiety. This is a well-validated scale with few somatic symptom items that can confound mood/anxiety assessment in medically-ill patients (Range: 0-21). Higher scores indicate higher levels of anxiety.
Change in Motivation to change | Baseline, 10-Week Follow-Up, 24-Week Follow-Up
  The University of Rhode Island Change Assessment (URICA) is a well-validated, 32-item measure that will be used to assess motivation to change. Higher scores indicate higher motivation to change.
Change in Exercise Identity | Baseline, 10-Week Follow-Up, 24-Week Follow-Up
  The Exercise Identity Scale (EIS) is a well-validated, 9-item measure that will be used to assess exercise identity (Range: 9-63). Higher scores indicate stronger exercise identity.
Change in General Self-Efficacy | Baseline, 10-Week Follow-Up, 24-Week Follow-Up
  Self-efficacy will be measured using the General Self Efficacy scale (GSE), a validated measure of self-efficacy, given its links to improved adherence. Higher scores indicate greater self-efficacy.
Change in Exercise-specific Self-efficacy | Baseline, 10-Week Follow-Up, 24-Week Follow-Up
  Exercise-specific self-efficacy will be measured by the Self-Efficacy for Exercise scale (SEE), a validated scale which assesses self-efficacy for exercise (Range: 0-90). Higher scores indicate higher self-efficacy.
Change in Internalized Weight Bias | Baseline, 10-Week Follow-Up, 24-Week Follow-Up
  The Weight Bias Internalization Scale - Modified (WBIS-M) is a well-validated, 11-item measure that will be used to measure internalized weight bias (Range: 11-77). Higher scores indicate greater internalized weight bias.
Change in Body Image | Baseline, 10-Week Follow-Up, 24-Week Follow-Up
  Body image will be assessed using the Multidimensional Body-Self Relations Questionnaire (MBSRQ). Higher scores indicate better body image.
Change in Bariatric Surgery-specific Diet and Vitamin Adherence | Baseline, 10-Week Follow-Up, 24-Week Follow-Up
  The Bariatric Surgery Self-Management Questionnaire (BSSQ) is a validated measure that will be used to assess adherence to diet and vitamin recommendations after bariatric surgery. Higher scores indicate better adherence to diet and vitamin recommendations.
Change in Self-Reported Physical Activity | Baseline, 10-Week Follow-Up, 24-Week Follow-Up
  The International Physical Activity Questionnaire (IPAQ) - Short Form is a well-validated 7-day physical activity recall assessment for physical activity. Activity will be measured by the number of MET-minutes of moderate or greater activity per week.
Change in Body weight | Baseline, 10-Week Follow-Up, 24-Week Follow-Up
  Body weight (in kilograms) will be measured on a calibrated scale.
Change in Waist circumference (in centimeters) | Baseline, 10-Week Follow-Up, 24-Week Follow-Up
  Waist circumference will be measured by a nurse.
Change in Blood pressure (millimeters of mercury) | Baseline, 10-Week Follow-Up, 24-Week Follow-Up
  Blood pressure will be measured by a nurse.
Change in Aerobic capacity and endurance | Baseline, 10-Week Follow-Up, 24-Week Follow-Up
  The 6 Minute Walk Test is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity.
Change in Social support for exercise | Baseline, 10-Week Follow-Up, 24-Week Follow-Up
  The Social Support and Exercise Survey is a 13-item validated measure that assesses social support for exercising from family and friends over the past 3 months. Scores range from 13 to 104, with higher scores indicating more social support.
Change in Social support for eating habits | Baseline, 10-Week Follow-Up, 24-Week Follow-Up
  The Social Support and Eating Habits Survey is a 10-item validated measure that assesses social support for healthy eating from family and friends over the past 3 months. Scores range from 10 to 80, with higher scores indicating more social support.
Change in Body composition | Baseline, 10-Week Follow-Up, 24-Week Follow-Up
  The measurement of body fat in relation to lean body mass will be measured using bio-electrical impedance.
Change in A1C | Baseline, 10-Week Follow-Up, 24-Week Follow-Up
  Hemoglobin A1C will be measured via blood draw.
Change in Lipids | Baseline, 10-Week Follow-Up, 24-Week Follow-Up
  Lipids will be measured via blood draw.
Change in Inflammation | Baseline, 10-Week Follow-Up, 24-Week Follow-Up
  C-reactive protein will be measured via blood draw as a measure of inflammation.
Change in Physical activity enjoyment | Baseline, 10-Week Follow-Up, 24-Week Follow-Up
  Self-efficacy will be measured using the Physical Activity Enjoyment Scale (PACES), a validated measure of enjoyment during exercise. Higher scores indicate greater enjoyment during exercise.

CONTACTS AND LOCATIONS:
Overall Officials: Emily H Feig, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Feig EH, Harnedy LE, Thorndike AN, Psaros C, Healy BC, Huffman JC. A Positive Emotion-Focused Intervention to Increase Physical Activity After Bariatric Surgery: Protocol for a Pilot Randomized Controlled Trial. JMIR Res Protoc. 2022 Oct 6;11(10):e39856. doi: 10.2196/39856. PMID 36201380